CLINICAL TRIAL: NCT01177046
Title: Development of a Multi-attribute Health Index to Measure the Quality of Labour Analgesia: Psychometric Development of a Quality of Neuraxial Labour Analgesia Scale
Brief Title: Development of a Multi-attribute Health Index: to Measure the Quality of Labour Analgesia: The QLA Index
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Pamela Angle, Anesthesiologist, Sunnybrook Health Sciences Centre
Other Study IDs: 160-2002
Record Dates: First submitted 2010-08-04; First posted 2010-08-06 (Estimated); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Labour Pain
Keywords: Women receiving labour epidural for most recent delivery
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The findings of this research will be used to develop a scale for measuring the quality of epidural pain relief achieved during labour and vaginal delivery.

DETAILED DESCRIPTION:
The current lack of a tool to measure the overall quality of neuraxial pain relief provided in labour analgesia trials has produced studies unable to provide clear direction to clinical care and research. Our previous work explored and described the underlying dimensions and attributes of quality neuraxial analgesia from the perspectives of labouring women as the initial phase of development of an Index to measure this as an outcome in research. We now seek to confirm our findings as well as to generate additional items (descriptors) of quality neuraxial analgesia from the perspectives of parturients and experts (obstetrical anesthesiologists and experienced labour nurses). Once generated, the full list of items will be used to in a subsequent study involving only parturients (Item Reduction phase) to develop a scale permitting global measurement of quality neuraxial labour analgesia. The resulting scale, once validated, will provide researchers with a simple global measure for quality in labour analgesia research. This scale will be used later in our program of research to assist with validation studies of the larger Multi-attribute Health Index we are developing.

ELIGIBILITY:
Inclusion Criteria:

1. Use of neuraxial labour analgesia during the current pregnancy
2. Native English-speakers
3. Term pregnancies (>37-42weeks)
4. The ability to read and write in English
5. Provision of written informed consent.

Exclusion Criteria:

1. Women who received IM or IV narcotics within 4 hours of epidural/ combined spinal epidural (CSE) placement
2. Women with evidence or history of maternal cognitive impairment
3. Women who experienced a neonatal death during the current pregnancy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women who received neuraxial labour analgesia during the current pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 752 (Actual)
Dates: Start 2010-07; Primary Completion 2021-10 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Psychometric instrument development study | 5-6 years
  Exploration and description of language, nature, and variability of women's pain experiences during labour and delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Pamela Angle, MD, MSc, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada